CLINICAL TRIAL: NCT06003777
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED, CROSSOVER, FIRST-IN-HUMAN STUDY TO ASSESS THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF SINGLE ASCENDING ORAL DOSES OF PF-06954522 IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Learn How Different Amounts of the Study Medicine Called PF-06954522 Are Tolerated and Act in the Body in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: C4001001; NCT06003777 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-08-03; First posted 2023-08-22 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Single dose administration of PF-06954522 and placebo. Participants will receive up to 5 dose levels of PF-06954522 and up to 2 dose levels of matching placebo.
  Interventions: Drug: PF-06954522; Drug: Placebo
- Cohort 2 (Experimental): Single dose administration of PF-06954522 and placebo. Participants will receive up to 4 dose levels of PF-06954522 and up to 2 dose levels of matching placebo.
  Interventions: Drug: PF-06954522; Drug: Placebo
- Cohort 3 (Experimental): Single dose administration of PF-06954522 and placebo. Participants will receive up to 2 dose levels of PF-06954522 and up to 1 dose level of matching placebo.
  Interventions: Drug: PF-06954522; Drug: Placebo

INTERVENTIONS:
Drug: PF-06954522 — PF-06954522 will be administered as oral suspensions as escalating single doses to be determined.
Drug: Placebo — Placebo will be administered as oral suspensions as escalating single doses to be determined.

SUMMARY:
The purposes of this study are:

* To see how the new medicine (PF-06954522) under study behave. And if there are any important side effects. A side effect is a reaction (expected or unexpected) to a medicine or treatment you take. The study will see how people feel after taking single increasing amount of the medicine by mouth.
* To measure the amount of study medicine in your blood after the medicine is taken by mouth.

This study is seeking for participants who:

* are females of 18 to 65 years old and are not able to give birth to a child.
* are males of 18 to 65 years old.
* have body mass index of 16 to 31 kilograms per meter squared.
* have a total body weight of more than 50 kilograms (110 pounds).

Participants will be chosen by chance, like drawing names out of a hat to receive either:

* study medicine (PF-06954522)
* or placebo (a pill that has no medicine in it).

Participants may receive up to 4 amounts of study medicine and up to 2 amounts of placebo. The time frame of the study is approximately up to 36 days for each group and participants will stay at CRU for 20 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants of non-childbearing potential aged 18 to 65 years, inclusive, at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
2. BMI of 16 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention, with the exception of moderate or strong cytochrome P450 3A (CYP3A) inducers or inhibitors which are prohibited within 14 days plus 5 half-lives prior to the first dose of study intervention.
3. Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer). Participation in studies of other investigational products (drug or vaccine) at any time during their participation in this study.
4. Standard 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results
5. Renal impairment as defined by an estimated glomerular filtration rate (eGFR) of <75 mL/min/1.73 m².
6. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

   * Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or bilirubin

     * 1.05 × upper limit of normal (ULN);
   * TSH > ULN;
   * HbA1c ≥6.5%;
   * Hematuria as defined by ≥1+ heme on urine dipstick;
   * Albuminuria as defined by urine albumin/creatinine ratio (UACR) >30 mg/g.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4001001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 26 participants (initially randomized participants and replacement participants) were enrolled in this study. All participants received at least 1 dose of study intervention and were assigned in the study into 3 cohorts. As planned, there were "replacement" participants in the study who may or may not be required to complete all periods of the cohort in which they were participating at the discretion of the principal investigator and sponsor.
Pre-assignment Details: In this study, dose have been reported from dose levels A to F, wherein Dose A is the lowest dose and Dose F is the highest dose received by study participants.
Groups:
- Cohort 1: Sequence 1: Participants received PF-06954522 matching placebo on Day 1 Period 1 then PF-06954522 dose level D in Period 2 then PF-06954522 dose level E in Period 3, PF-06954522 dose level D fed state high fat in Period 4 followed by PF-06954522 dose level F in Period 5. There was a washout period of 7 days in between each period.
- Cohort 1: Sequence 2: Participants received PF-06954522 dose level C on Day 1 Period 1 then PF-06954522 matching placebo in Period 2 then PF-06954522 dose level E in Period 3, PF-06954522 matching placebo in Period 4 in fed state (high-fat meal) followed by PF-06954522 dose level F in Period 5. There was a washout period of 7 days in between each period.
- Cohort 1: Sequence 3: Participants received PF-06954522 dose level C on Day 1 Period 1 then PF-06954522 dose level D in Period 2 then PF-06954522 matching placebo in Period 3, PF-06954522 dose level D fed state high fat in Period 4 followed by PF-06954522 dose level F in Period 5. There was a washout period of 7 days in between each period.
- Cohort 1: Sequence 4: Participants received PF-06954522 dose level C on Day 1 Period 1 then PF-06954522 dose level D in Period 2 then PF-06954522 dose level E in Period 3, PF-06954522 dose level D in Period 4 in fed state (high-fat meal) followed by PF-06954522 matching placebo in Period 5. There was a washout period of 7 days in between each period.
- Cohort 1: Sequence 5: Participants received PF-06954522 dose level C on Day 1 Period 1 then PF-06954522 dose level D in Period 2 then PF-06954522 dose level E in Period 3, PF-06954522 dose level D fed state high fat in Period 4 followed by PF-06954522 dose level F in Period 5. There was a washout period of 7 days in between each period.
- Cohort 2: Sequence 1: Participants received PF-06954522 matching placebo on Day 1 Period 1 then PF-06954522 dose level A fed state standard meal in Period 2 then PF-06954522 dose level B fed state high fat meal in Period 3 followed by PF-06954522 dose level F in Period 4. There was a washout period of 7 days in between each period.
- Cohort 2: Sequence 2: Participants received PF-06954522 dose level B on Day 1 Period 1 then PF-06954522 matching placebo in Period 2 in fed state (standard meal) then PF-06954522 matching placebo in Period 3 in fed state (high-fat meal) followed by PF-06954522 dose level F in Period 4. There was a washout period of 7 days in between each period.
- Cohort 2: Sequence 3: Participants received PF-06954522 dose level B on Day 1 Period 1 then PF-06954522 dose level A fed state standard meal in Period 2 then PF-06954522 dose level B fed state high fat in Period 3 followed by PF-06954522 dose level F in Period 4. There was a washout period of 7 days in between each period.
- Cohort 2: Sequence 4: Participants received PF-06954522 dose level B on Day 1 Period 1 then PF-06954522 dose level A fed state standard meal in Period 2 then PF-06954522 dose level B fed state high fat in Period 3 followed by PF-06954522 matching placebo in Period 4. There was a washout period of 7 days in between each period.
- Cohort 3: Sequence 1: Japanese participants received PF-06954522 matching placebo on Day 1 Period 1 then PF-06954522 dose level E in Period 2 followed by PF-06954522 matching placebo in Period 3 in fed state (high-fat meal). There was a washout period of 7 days in between each period.
- Cohort 3: Sequence 2: Japanese participants received PF-06954522 dose level D on Day 1 Period 1 then PF-06954522 matching placebo in Period 2 followed by PF-06954522 dose level D fed state high fat in Period 3. There was a washout period of 7 days in between each period.
- Cohort 3: Sequence 3: Japanese participants received PF-06954522 dose level D on Day 1 Period 1 then PF-06954522 dose level E in Period 2 followed by PF-06954522 dose level D fed state high fat in Period 3. There was a washout period of 7 days in between each period.
Period: Period 1
Arm/Group | Cohort 1: Sequence 1 | Cohort 1: Sequence 2 | Cohort 1: Sequence 3 | Cohort 1: Sequence 4 | Cohort 1: Sequence 5 | Cohort 2: Sequence 1 | Cohort 2: Sequence 2 | Cohort 2: Sequence 3 | Cohort 2: Sequence 4 | Cohort 3: Sequence 1 | Cohort 3: Sequence 2 | Cohort 3: Sequence 3
Started | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 1 | 1 | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Cohort 1: Sequence 1 | Cohort 1: Sequence 2 | Cohort 1: Sequence 3 | Cohort 1: Sequence 4 | Cohort 1: Sequence 5 | Cohort 2: Sequence 1 | Cohort 2: Sequence 2 | Cohort 2: Sequence 3 | Cohort 2: Sequence 4 | Cohort 3: Sequence 1 | Cohort 3: Sequence 2 | Cohort 3: Sequence 3
Started | 2 | 2 (Participants may not have taken part in all study periods (including, for example, replacement participants). Therefore, the number of participants starting a period may not be equal to the number completing the previous period.) | 2 (Participants may not have taken part in all study periods (including, for example, replacement participants). Therefore, the number of participants starting a period may not be equal to the number completing the previous period.) | 2 | 2 (Participants may not have taken part in all study periods (including, for example, replacement participants). Therefore, the number of participants starting a period may not be equal to the number completing the previous period.) | 2 | 2 | 2 | 2 | 2 | 2 | 1 (Participants may not have taken part in all study periods (including, for example, replacement participants). Therefore, the number of participants starting a period may not be equal to the number completing the previous period.)
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Period 3
Arm/Group | Cohort 1: Sequence 1 | Cohort 1: Sequence 2 | Cohort 1: Sequence 3 | Cohort 1: Sequence 4 | Cohort 1: Sequence 5 | Cohort 2: Sequence 1 | Cohort 2: Sequence 2 | Cohort 2: Sequence 3 | Cohort 2: Sequence 4 | Cohort 3: Sequence 1 | Cohort 3: Sequence 2 | Cohort 3: Sequence 3
Started | 2 | 2 | 2 | 2 | 2 | 1 (Participants may not have taken part in all study periods (including, for example, replacement participants). Therefore, the number of participants starting a period may not be equal to the number completing the previous period.) | 2 | 2 | 1 | 2 | 2 | 2 (Participants may not have taken part in all study periods (including, for example, replacement participants). Therefore, the number of participants starting a period may not be equal to the number completing the previous period.)
Completed | 2 | 2 | 2 | 2 | 2 | 1 | 1 | 2 | 1 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Cohort 1: Sequence 1 | Cohort 1: Sequence 2 | Cohort 1: Sequence 3 | Cohort 1: Sequence 4 | Cohort 1: Sequence 5 | Cohort 2: Sequence 1 | Cohort 2: Sequence 2 | Cohort 2: Sequence 3 | Cohort 2: Sequence 4 | Cohort 3: Sequence 1 | Cohort 3: Sequence 2 | Cohort 3: Sequence 3
Started | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 1 | 0 (There was no period 4 in cohort 3.) | 0 (There was no period 4 in cohort 3.) | 0 (There was no period 4 in cohort 3.)
Completed | 2 | 1 | 1 | 2 | 2 | 2 | 1 | 2 | 1 | 0 | 0 | 0
Not Completed | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — No longer met eligibility criteria | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | Cohort 1: Sequence 1 | Cohort 1: Sequence 2 | Cohort 1: Sequence 3 | Cohort 1: Sequence 4 | Cohort 1: Sequence 5 | Cohort 2: Sequence 1 | Cohort 2: Sequence 2 | Cohort 2: Sequence 3 | Cohort 2: Sequence 4 | Cohort 3: Sequence 1 | Cohort 3: Sequence 2 | Cohort 3: Sequence 3
Started | 2 | 1 | 1 | 2 | 2 | 0 (There was no period 5 in cohort 2 or 3.) | 0 (There was no period 5 in cohort 2 or 3.) | 0 (There was no period 5 in cohort 2 or 3.) | 0 (There was no period 5 in cohort 2 or 3.) | 0 (There was no period 5 in cohort 2 or 3.) | 0 (There was no period 5 in cohort 2 or 3.) | 0 (There was no period 5 in cohort 2 or 3.)
Completed | 2 | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants randomly assigned to study intervention and who received at least 1 dose of study intervention. Data for baseline characteristics provided per cohort as prespecified in statistical analysis plan.
Groups:
- Cohort 1: Participants received up to 5 dose levels of PF-06954522 and matching placebo.
- Cohort 2: Participants received up to 4 dose levels of PF-06954522 and matching placebo.
- Cohort 3: Participants received up to 3 dose levels of PF-06954522 and matching placebo.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 12 | 8 | 6 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.6 (9.84) | 42.1 (11.44) | 42.5 (12.28) | 42.9 (10.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 0 | 3
  Male | 9 | 8 | 6 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 0 | 10
  Not Hispanic or Latino | 7 | 3 | 6 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 6 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 0 | 7
  White | 7 | 3 | 0 | 10
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AEs) was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE was considered a TEAE if the event started during the effective duration of treatment. All events that start on or after the first dose of study intervention, but before the end of the study were flagged as TEAEs. Serious AE (SAE) was defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria: death, life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly or birth defect. AEs included SAEs and non-SAEs.
Time Frame: From Day 1 up to 35 days after last of study drug (maximum up to approximately 88 days)
Population: Safety analysis set included all participants randomly assigned to study intervention and who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: PF-06954522 Dose Level C: Participants received PF-06954522 dose level C in fasted state.
- Cohort 1: PF-06954522 Dose Level D: Participants received PF-06954522 dose level D in fasted state.
- Cohort 1: PF-06954522 Dose Level D (Fed State High Fat Meal): Participants received PF-06954522 dose level D in fed state with a high fat meal.
- Cohort 1: PF-06954522 Dose Level E: Participants received PF-06954522 dose level E in fasted state.
- Cohort 1: PF-06954522 Dose Level F: Participants received PF-06954522 dose level F in fasted state.
- Cohort 1 and 2: Placebo (Fasted State): Participants received PF-06954522 matching placebo in fasted state.
- Cohort 1 and 2: Placebo (Fed State): Participants received PF-06954522 matching placebo in fed state with high fat meal.
Arm/Group | Cohort 1: PF-06954522 Dose Level C | Cohort 1: PF-06954522 Dose Level D | Cohort 1: PF-06954522 Dose Level D (Fed State High Fat Meal) | Cohort 1: PF-06954522 Dose Level E | Cohort 1: PF-06954522 Dose Level F | Cohort 1 and 2: Placebo (Fasted State) | Cohort 1 and 2: Placebo (Fed State)
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 6 | 11 | 4
Participants | 5 | 8 | 6 | 8 | 6 | 3 | 1

2. Primary Outcome: Cohort 2: Number of Participants With TEAEs
Description: An AEs was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE was considered a TEAE if the event started during the effective duration of treatment. All events that start on or after the first dose of study intervention, but before the end of the study were flagged as TEAEs. SAE was defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria: death, life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly or birth defect. AEs included SAEs and non-SAEs.
Time Frame: From Day 1 up to 35 days after last of study drug (maximum up to approximately 76 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: Placebo (Fed-standard Meal): Participants received PF-06954522 matching placebo in the fed state standard-meal.
- Cohort 1 and 2: Placebo (Fed-high Fat Meal): Participants received PF-06954522 matching placebo in the fed state high-fat meal.
- Cohort 2: PF-06954522 Dose Level A (Fed State-standard Meal): Participants received PF-06954522 dose level A in the fed state standard-meal.
- Cohort 2: PF-06954522 Dose Level B: Participants received PF-06954522 dose level B in fasted state.
- Cohort 2: PF-06954522 Dose Level B (Fed State High-fat Meal): Participants received PF-06954522 dose level B in the fed state high-fat meal.
- Cohort 2: PF-06954522 Dose Level F: Participants received PF-06954522 dose level F in fasted state.
Arm/Group | Cohort 1 and 2: Placebo (Fasted State) | Cohort 2: Placebo (Fed-standard Meal) | Cohort 1 and 2: Placebo (Fed-high Fat Meal) | Cohort 2: PF-06954522 Dose Level A (Fed State-standard Meal) | Cohort 2: PF-06954522 Dose Level B | Cohort 2: PF-06954522 Dose Level B (Fed State High-fat Meal) | Cohort 2: PF-06954522 Dose Level F
Number analyzed (Participants) | 11 | 2 | 4 | 6 | 6 | 4 | 5
Participants | 3 | 0 | 1 | 2 | 2 | 0 | 5

3. Primary Outcome: Cohort 3: Number of Participants With TEAEs
Description: as for outcome 2
Time Frame: From Day 1 up to 35 days after last of study drug (maximum up to approximately 64 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 3: Placebo: Japanese participants received a single dose of matching placebo to PF-06954522 on Day 1 of Cohort 3.
- Cohort 3: Placebo (Fed): Japanese participants received a single dose of matching placebo to PF-06954522 in the fed state high-fat meal on Day 1 of Cohort 3.
- Cohort 3: PF-06954522 Dose Level D: Japanese participants received PF-06954522 dose level D on Day 1 of Cohort 3.
- Cohort 3: PF-06954522 Dose Level D (Fed State High-fat Meal): Japanese participants received PF-06954522 dose level D in the fed state high-fat meal on Day 1 of Cohort 3.
- Cohort 3: PF-06954522 Dose Level E: Japanese participants received PF-06954522 dose level E on Day 1 of Cohort 3.
Arm/Group | Cohort 3: Placebo | Cohort 3: Placebo (Fed) | Cohort 3: PF-06954522 Dose Level D | Cohort 3: PF-06954522 Dose Level D (Fed State High-fat Meal) | Cohort 3: PF-06954522 Dose Level E
Number analyzed (Participants) | 4 | 2 | 4 | 4 | 3
Participants | 3 | 2 | 4 | 4 | 3

4. Primary Outcome: Cohort 1: Number of Participants With Hematology Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: Planned hematology laboratory tests included: hematocrit, red blood cell count, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils and lymphocytes. The number of participants with results meeting pre-specified criteria (without regard to baseline abnormality) is reported.
Time Frame: From Day 1 up to 35 days after last of study drug (maximum up to approximately 88 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: PF-06954522 Dose Level D (Fed State High Fat Meal: Participants received PF-06954522 dose level D in fed state with a high fat meal.
- Cohort 1 and 2: Placebo (Fed State): Participants received PF-06954522 matching placebo in fed state high fat meal.
Arm/Group | Cohort 1: PF-06954522 Dose Level C | Cohort 1: PF-06954522 Dose Level D | Cohort 1: PF-06954522 Dose Level D (Fed State High Fat Meal | Cohort 1: PF-06954522 Dose Level E | Cohort 1: PF-06954522 Dose Level F | Cohort 1 and 2: Placebo (Fasted State) | Cohort 1 and 2: Placebo (Fed State)
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 6 | 11 | 4
Participants | 0 | 0 | 3 | 2 | 1 | 3 | 2

5. Primary Outcome: Cohort 2: Number of Participants With Hematology Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: as for outcome 4
Time Frame: From Day 1 up to 35 days after last of study drug (maximum up to approximately 76 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: Placebo (Fed-standard Meal): Participants received PF-06954522 matching placebo in the fed standard-meal state.
Arm/Group | Cohort 1 and 2: Placebo (Fasted State) | Cohort 2: Placebo (Fed-standard Meal) | Cohort 1 and 2: Placebo (Fed-high Fat Meal) | Cohort 2: PF-06954522 Dose Level A (Fed State-standard Meal) | Cohort 2: PF-06954522 Dose Level B | Cohort 2: PF-06954522 Dose Level B (Fed State High-fat Meal) | Cohort 2: PF-06954522 Dose Level F
Number analyzed (Participants) | 11 | 2 | 4 | 6 | 6 | 4 | 5
Participants | 3 | 1 | 2 | 3 | 2 | 1 | 4

6. Primary Outcome: Cohort 3: Number of Participants With Hematology Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: as for outcome 4
Time Frame: From Day 1 up to 35 days after last of study drug (maximum up to approximately 64 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: Placebo (Fed) | Cohort 3: PF-06954522 Dose Level D | Cohort 3: PF-06954522 Dose Level D (Fed State High-fat Meal) | Cohort 3: PF-06954522 Dose Level E
Number analyzed (Participants) | 4 | 2 | 4 | 4 | 3
Participants | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Cohort 1: Number of Participants With Clinical Chemistry Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: Planned chemistry laboratory tests included: blood urea nitrogen, creatinine, cystatin C, estimated glomerular filtration rate, glucose (fasting), calcium, sodium, potassium. chloride, total bicarbonate, aspartate aminotransferase, alanine aminotransferase, total bilirubin, direct and indirect bilirubin, gamma-glutamyl transferase, alkaline phosphatase, creatine kinase, uric acid, albumin and total protein. The number of participants with results meeting pre-specified criteria (without regard to baseline abnormality) is reported.
Time Frame: From Day 1 up to 35 days after last of study drug (maximum up to approximately 88 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-06954522 Dose Level C | Cohort 1: PF-06954522 Dose Level D | Cohort 1: PF-06954522 Dose Level D (Fed State High Fat Meal) | Cohort 1: PF-06954522 Dose Level E | Cohort 1: PF-06954522 Dose Level F | Cohort 1 and 2: Placebo (Fasted State) | Cohort 1 and 2: Placebo (Fed State)
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 6 | 11 | 4
Participants | 0 | 0 | 0 | 2 | 0 | 3 | 0

8. Primary Outcome: Cohort 2: Number of Participants With Clinical Chemistry Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: as for outcome 7
Time Frame: From Day 1 up to 35 days after last of study drug (maximum up to approximately 76 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 and 2: Placebo (Fasted State) | Cohort 2: Placebo (Fed-standard Meal) | Cohort 1 and 2: Placebo (Fed-high Fat Meal) | Cohort 2: PF-06954522 Dose Level A (Fed State-standard Meal) | Cohort 2: PF-06954522 Dose Level B | Cohort 2: PF-06954522 Dose Level B (Fed State High-fat Meal) | Cohort 2: PF-06954522 Dose Level F
Number analyzed (Participants) | 11 | 2 | 4 | 6 | 6 | 4 | 5
Participants | 3 | 0 | 0 | 2 | 1 | 0 | 2

9. Primary Outcome: Cohort 3: Number of Participants With Clinical Chemistry Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: as for outcome 7
Time Frame: From Day 1 up to 35 days after last of study drug (maximum up to approximately 64 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: Placebo (Fed) | Cohort 3: PF-06954522 Dose Level D | Cohort 3: PF-06954522 Dose Level D (Fed State High-fat Meal) | Cohort 3: PF-06954522 Dose Level E
Number analyzed (Participants) | 4 | 2 | 4 | 4 | 3
Participants | 1 | 0 | 1 | 1 | 0

10. Primary Outcome: Cohort 1: Number of Participants With Urinalysis Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: Planned urinalysis laboratory tests included: pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, urobilinogen and urine bilirubin. The number of participants with results meeting pre-specified criteria (without regard to baseline abnormality) is reported.
Time Frame: From Day 1 up to 35 days after last of study drug (maximum up to approximately 88 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-06954522 Dose Level C | Cohort 1: PF-06954522 Dose Level D | Cohort 1: PF-06954522 Dose Level D (Fed State High Fat Meal) | Cohort 1: PF-06954522 Dose Level E | Cohort 1: PF-06954522 Dose Level F | Cohort 1 and 2: Placebo (Fasted State) | Cohort 1 and 2: Placebo (Fed State)
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 6 | 11 | 4
Participants | 2 | 3 | 6 | 3 | 3 | 5 | 2

11. Primary Outcome: Cohort 2: Number of Participants With Urinalysis Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: as for outcome 10
Time Frame: From Day 1 up to 35 days after last of study drug (maximum up to approximately 76 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 and 2: Placebo (Fasted State) | Cohort 2: Placebo (Fed-standard Meal) | Cohort 1 and 2: Placebo (Fed-high Fat Meal) | Cohort 2: PF-06954522 Dose Level A (Fed State-standard Meal) | Cohort 2: PF-06954522 Dose Level B | Cohort 2: PF-06954522 Dose Level B (Fed State High-fat Meal) | Cohort 2: PF-06954522 Dose Level F
Number analyzed (Participants) | 11 | 2 | 4 | 6 | 6 | 4 | 5
Participants | 5 | 1 | 2 | 2 | 5 | 1 | 3

12. Primary Outcome: Cohort 3: Number of Participants With Urinalysis Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: as for outcome 10
Time Frame: From Day 1 up to 35 days after last of study drug (maximum up to approximately 64 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: Placebo (Fed) | Cohort 3: PF-06954522 Dose Level D | Cohort 3: PF-06954522 Dose Level D (Fed State High-fat Meal) | Cohort 3: PF-06954522 Dose Level E
Number analyzed (Participants) | 4 | 2 | 4 | 4 | 3
Participants | 0 | 0 | 2 | 1 | 1

13. Primary Outcome: Cohort 1: Number of Participants According to Categorization of Vital Signs Abnormalities Data
Description: Vital signs parameters were summarized according to pre-specified categorization of data: supine systolic blood pressure: Value less than (<) 90 millimeter of mercury (mmHg), increase or decrease from baseline >= 30mmHg, supine diastolic blood pressure: value <50 mmHg, increase or decrease from baseline >= 20mmHg and supine pulse rate: Value < 40 beats per minute bpm or > 120bpm.
Time Frame: From Day 1 up to 35 days after last of study drug (maximum up to approximately 88 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-06954522 Dose Level C | Cohort 1: PF-06954522 Dose Level D | Cohort 1: PF-06954522 Dose Level D (Fed State High Fat Meal) | Cohort 1: PF-06954522 Dose Level E | Cohort 1: PF-06954522 Dose Level F | Cohort 1 and 2: Placebo (Fasted State) | Cohort 1 and 2: Placebo (Fed State)
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 6 | 11 | 4
Participants
  Supine systolic blood pressure: Value < 90mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine systolic blood pressure : Increase from baseline >= 30mmHg | 1 | 1 | 0 | 3 | 1 | 0 | 0
  Supine diastolic blood pressure: Increase from baseline >= 20mmHg | 0 | 3 | 0 | 4 | 0 | 0 | 0
  Supine pulse rate: Value > 120bpm | 0 | 0 | 0 | 1 | 0 | 0 | 0

14. Primary Outcome: Cohort 2: Number of Participants According to Categorization of Vital Signs Abnormalities Data
Description: as for outcome 13
Time Frame: From Day 1 up to 35 days after last of study drug (maximum up to approximately 76 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 and 2: Placebo (Fasted State) | Cohort 2: Placebo (Fed-standard Meal) | Cohort 1 and 2: Placebo (Fed-high Fat Meal) | Cohort 2: PF-06954522 Dose Level A (Fed State-standard Meal) | Cohort 2: PF-06954522 Dose Level B | Cohort 2: PF-06954522 Dose Level B (Fed State High-fat Meal) | Cohort 2: PF-06954522 Dose Level F
Number analyzed (Participants) | 11 | 2 | 4 | 6 | 6 | 4 | 5
Participants
  Supine systolic blood pressure: Value < 90mmHg | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Supine systolic blood pressure : Increase from baseline >= 30mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Supine diastolic blood pressure: Increase from baseline >= 20mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Supine pulse rate: Value > 120bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: Cohort 3: Number of Participants According to Categorization of Vital Signs Abnormalities Data
Description: Vital signs parameters were summarized according to pre-specified categorization of data: supine systolic blood pressure: Value less than (<) 90 millimeter of mercury (mmHg), increase or decrease from baseline >= 30mmHg, supine diastolic blood pressure: value <50 mmHg and increase or decrease from baseline >= 20mmHg.
Time Frame: From Day 1 up to 35 days after last of study drug (maximum up to approximately 64 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: Placebo (Fed) | Cohort 3: PF-06954522 Dose Level D | Cohort 3: PF-06954522 Dose Level D (Fed State High-fat Meal) | Cohort 3: PF-06954522 Dose Level E
Number analyzed (Participants) | 4 | 2 | 4 | 4 | 3
Participants
  Supine systolic blood pressure: Value < 90mmHg | 0 | 0 | 1 | 0 | 1
  Supine systolic blood pressure : Increase from baseline >= 30mmHg | 0 | 0 | 1 | 0 | 2
  Supine diastolic blood pressure: Increase from baseline >= 20mmHg | 0 | 0 | 1 | 0 | 1

16. Primary Outcome: Cohort 1: Number of Participants According to Categorization of Electrocardiogram (ECG) Abnormalities Parameters
Description: Pre-specified ECG abnormalities criteria : PR interval millisecond (msec), value >=300, baseline > 200 and percentage (%) change >=25%, baseline <=200 and percentage change >=50%; QRS duration (msec): value >=140, % change>= 50%; corrected QT interval using Fridericia's formula (QTcF) (msec): 450 < value <= 480, 480<= value <500, value >=500, 30<= change <60 and change > 60.
Time Frame: From Day 1 up to 35 days after last of study drug (maximum up to approximately 88 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-06954522 Dose Level C | Cohort 1: PF-06954522 Dose Level D | Cohort 1: PF-06954522 Dose Level D (Fed State High Fat Meal) | Cohort 1: PF-06954522 Dose Level E | Cohort 1: PF-06954522 Dose Level F | Cohort 1 and 2: Placebo (Fasted State) | Cohort 1 and 2: Placebo (Fed State)
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 6 | 11 | 4
Participants
  PR interval: value >=300 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR interval: baseline > 200 and % change >=25% | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR interval: baseline <=200 and percentage change >=50% | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS duration: value >=140 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS duration: % change>= 50% | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF: 450 < value <= 480 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  QTcF: 480<= value <500 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF: value >=500 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF: 30<= change <60 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF: change >60 | 0 | 0 | 1 | 0 | 0 | 0 | 0

17. Primary Outcome: Cohort 2: Number of Participants According to Categorization of ECG Abnormalities Parameters
Description: as for outcome 16
Time Frame: From Day 1 up to 35 days after last of study drug (maximum up to approximately 76 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 and 2: Placebo (Fasted State) | Cohort 2: Placebo (Fed-standard Meal) | Cohort 1 and 2: Placebo (Fed-high Fat Meal) | Cohort 2: PF-06954522 Dose Level A (Fed State-standard Meal) | Cohort 2: PF-06954522 Dose Level B | Cohort 2: PF-06954522 Dose Level B (Fed State High-fat Meal) | Cohort 2: PF-06954522 Dose Level F
Number analyzed (Participants) | 11 | 2 | 4 | 6 | 6 | 4 | 5
Participants
  PR interval: value >=300 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR interval: baseline > 200 and % change >=25% | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR interval: baseline <=200 and percentage change >=50% | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS duration: value >=140 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS duration: % change>= 50% | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF: 450 < value <= 480 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF: 480<= value <500 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF: value >=500 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF: 30<= change <60 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF: change >60 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Primary Outcome: Cohort 3: Number of Participants According to Categorization of ECG Abnormalities Parameters
Description: as for outcome 16
Time Frame: From Day 1 up to 35 days after last of study drug (maximum up to approximately 64 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: Placebo (Fed) | Cohort 3: PF-06954522 Dose Level D | Cohort 3: PF-06954522 Dose Level D (Fed State High-fat Meal) | Cohort 3: PF-06954522 Dose Level E
Number analyzed (Participants) | 4 | 2 | 4 | 4 | 3
Participants
  PR interval: value >=300 | 0 | 0 | 0 | 0 | 0
  PR interval: baseline > 200 and % change >=25% | 0 | 0 | 0 | 0 | 0
  PR interval: baseline <=200 and percentage change >=50% | 0 | 0 | 0 | 0 | 0
  QRS duration: value >=140 | 0 | 0 | 0 | 0 | 0
  QRS duration: % change>= 50% | 0 | 0 | 0 | 0 | 0
  QTcF: 450 <value <=480 | 0 | 0 | 0 | 0 | 0
  QTcF: 480<= value <500 | 0 | 0 | 0 | 0 | 0
  QTcF: value >=500 | 0 | 0 | 0 | 0 | 0
  QTcF: 30<= change <60 | 0 | 0 | 0 | 0 | 0
  QTcF: change >60 msec | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Cohort 1: Area Under the Plasma Concentration-Time Profile From Time Zero (0) to Time of Last Quantifiable Concentration (AUClast) of PF-06954522
Description: AUClast was determined by using linear/log trapezoidal method.
Time Frame: From 0 hours (pre-dose) to 72 hours following a single dose on Day 1
Population: Pharmacokinetic (PK) parameter set included all participants who were randomly assigned to study intervention and received at least 1 dose of study intervention and had at least 1 of the PK parameters of interest calculated. Data for cohorts and periods included in the pre-specified secondary outcome measure are reported here (i.e., cohort 1, plasma concentration parameters observed following administration of PF-06954522 in the fasted state).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Cohort 1: PF-06954522 Dose Level C | Cohort 1: PF-06954522 Dose Level D | Cohort 1: PF-06954522 Dose Level E | Cohort 1: PF-06954522 Dose Level F
Number analyzed (Participants) | 7 | 8 | 8 | 6
Nanogram*hour per milliliter (ng*hr/mL) | 1394 (37) | 4252 (43) | 7503 (60) | 5631 (40)

20. Secondary Outcome: Cohort 2: AUClast of PF-06954522
Description: AUClast was determined by using linear/log trapezoidal method.
Time Frame: From 0 hours (pre-dose) to 72 hours following a single dose on Day 1
Population: PK parameter set included all participants who were randomly assigned to study intervention and received at least 1 dose of study intervention and had at least 1 of the PK parameters of interest calculated. Data for cohorts and periods included in the pre-specified secondary outcome measure are reported here (i.e., cohort 2, plasma concentration parameters observed following administration of PF-06954522 in the fasted state).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 2: PF-06954522 Dose Level B | Cohort 2: PF-06954522 Dose Level F
Number analyzed (Participants) | 6 | 5
ng*hr/mL | 827.2 (24) | 12630 (40)

21. Secondary Outcome: Cohort 1: Maximum Observed Concentration (Cmax) of PF-06954522
Description: Cmax of PF-06954522 was reported in this outcome measure.
Time Frame: From 0 hours (pre-dose) to 72 hours following a single dose on Day 1
Population: PK parameter set included all participants who were randomly assigned to study intervention and received at least 1 dose of study intervention and had at least 1 of the PK parameters of interest calculated. Data for cohorts and periods included in the pre-specified secondary outcome measure are reported here (i.e., cohort 1, plasma concentration parameters observed following administration of PF-06954522 in the fasted state).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1: PF-06954522 Dose Level C | Cohort 1: PF-06954522 Dose Level D | Cohort 1: PF-06954522 Dose Level E | Cohort 1: PF-06954522 Dose Level F
Number analyzed (Participants) | 7 | 8 | 8 | 6
Nanogram per milliliter (ng/mL) | 112.9 (40) | 377.7 (38) | 837.6 (53) | 522.9 (55)

22. Secondary Outcome: Cohort 2: Cmax of PF-06954522
Description: Cmax of PF-06954522 was reported in this outcome measure.
Time Frame: From 0 hours (pre-dose) to 72 hours following a single dose on Day 1
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 2: PF-06954522 Dose Level B | Cohort 2: PF-06954522 Dose Level F
Number analyzed (Participants) | 6 | 5
ng/mL | 86.82 (28) | 1088 (57)

23. Secondary Outcome: Cohort 1: Time to Maximum Observed Concentration (Tmax) of PF-06954522
Description: Tmax of PF-06954522 was reported in this outcome measure.
Time Frame: From 0 hours (pre-dose) to 72 hours following a single dose on Day 1
Population: as for outcome 21
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: PF-06954522 Dose Level C | Cohort 1: PF-06954522 Dose Level D | Cohort 1: PF-06954522 Dose Level E | Cohort 1: PF-06954522 Dose Level F
Number analyzed (Participants) | 7 | 8 | 8 | 6
Hours | 1.02 [1.00 to 2.00] | 3.00 [1.02 to 12.0] | 2.02 [1.00 to 6.00] | 1.09 [1.03 to 4.00]

24. Secondary Outcome: Cohort 2: Tmax of PF-06954522
Description: Tmax of PF-06954522 was reported in this outcome measure.
Time Frame: From 0 hours (pre-dose) to 72 hours following a single dose on Day 1
Population: as for outcome 20
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 2: PF-06954522 Dose Level B | Cohort 2: PF-06954522 Dose Level F
Number analyzed (Participants) | 6 | 5
Hours | 2.04 [1.00 to 4.05] | 1.00 [0.600 to 4.00]

25. Secondary Outcome: Cohort 1: Area Under the Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUCinf) of PF-06954522
Description: Area under the plasma concentration-time profile from time 0 extrapolated to infinite time. It was determined by AUClast +(Clast*/kel), where Clast is the predicted plasma concentration at the last quantifiable timepoint estimated from the log-linear regression analysis.
Time Frame: From 0 hours (pre-dose) to 72 hours following a single dose on Day 1
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter (ng.hr/mL)
Arm/Group | Cohort 1: PF-06954522 Dose Level C | Cohort 1: PF-06954522 Dose Level D | Cohort 1: PF-06954522 Dose Level E | Cohort 1: PF-06954522 Dose Level F
Number analyzed (Participants) | 7 | 8 | 8 | 6
Nanogram*hour per milliliter (ng.hr/mL) | 1415 (36) | 4283 (43) | 7576 (60) | 5667 (40)

26. Secondary Outcome: Cohort 2: AUCinf of PF-06954522
Description: as for outcome 25
Time Frame: From 0 hours (pre-dose) to 72 hours following a single dose on Day 1
Population: PK parameter set: all participants who were randomly assigned to study intervention & received at least 1 dose of study intervention & had at least 1 of PK parameters of interest calculated. "Overall Number of Participants Analyzed" signifies participants evaluable for this parameter. Data for cohorts and periods included in pre-specified secondary outcome measure are reported here (i.e., cohort 2, plasma concentration parameters observed following administration of PF-06954522 in fasted state).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hr/mL
Arm/Group | Cohort 2: PF-06954522 Dose Level B | Cohort 2: PF-06954522 Dose Level F
Number analyzed (Participants) | 6 | 5
ng.hr/mL | 846.6 (23) | 12700 (40)

27. Secondary Outcome: Cohort 1: Terminal Half-Life (t1/2) of PF-06954522
Description: t1/2 was determined by Loge (2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: From 0 hours (pre-dose) to 72 hours following a single dose on Day 1
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Cohort 1: PF-06954522 Dose Level C | Cohort 1: PF-06954522 Dose Level D | Cohort 1: PF-06954522 Dose Level E | Cohort 1: PF-06954522 Dose Level F
Number analyzed (Participants) | 7 | 8 | 8 | 6
Hours | 6.313 (1.4278) | 8.444 (3.3668) | 7.264 (2.8676) | 5.958 (1.6741)

28. Secondary Outcome: Cohort 2: t1/2 of PF-06954522
Description: t1/2was determined by Loge (2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: From 0 hours (pre-dose) to 72 hours following a single dose on Day 1
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Cohort 2: PF-06954522 Dose Level B | Cohort 2: PF-06954522 Dose Level F
Number analyzed (Participants) | 6 | 5
Hours | 5.918 (0.74714) | 7.766 (2.6585)

ADVERSE EVENTS:
Time Frame: From Day 1 to up to 35 days after last dose of study intervention (maximum up to 88 days for Cohort 1, 76 days for Cohort 2 and 64 days for Cohort 3)
Description: Same event may appear as both non-SAE and SAE but what is presented are distinct events. An event may be categorized as serious in one participant and non-serious in another participant or one participant may have experienced both serious and non-serious event. Safety analysis set included all participants who received at least one dose of investigational product.
Groups:
- Cohort 2: Placebo Standard Meal: Participants received PF-06954522 matching placebo in the standard meal.
- Cohort 3: Placebo: Japanese participants received a single dose of matching placebo of PF-06954522 on Day 1 of Cohort 3.
Arm/Group | Cohort 1 and 2: Placebo (Fasted State) | Cohort 1 and 2: Placebo (Fed State) | Cohort 1: PF-06954522 Dose Level C | Cohort 1: PF-06954522 Dose Level D | Cohort 1: PF-06954522 Dose Level D (Fed State High Fat Meal) | Cohort 1: PF-06954522 Dose Level E | Cohort 1: PF-06954522 Dose Level F | Cohort 2: Placebo Standard Meal | Cohort 2: PF-06954522 Dose Level A (Fed State-standard Meal) | Cohort 2: PF-06954522 Dose Level B | Cohort 2: PF-06954522 Dose Level B (Fed State High-fat Meal) | Cohort 2: PF-06954522 Dose Level F | Cohort 3: Placebo | Cohort 3: Placebo (Fed) | Cohort 3: PF-06954522 Dose Level D | Cohort 3: PF-06954522 Dose Level D (Fed State High-fat Meal) | Cohort 3: PF-06954522 Dose Level E
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/4 | 0/7 | 0/8 | 0/8 | 0/8 | 0/6 | 0/2 | 0/6 | 0/6 | 0/4 | 0/5 | 0/4 | 0/2 | 0/4 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/4 | 0/7 | 0/8 | 0/8 | 0/8 | 0/6 | 0/2 | 0/6 | 0/6 | 0/4 | 0/5 | 0/4 | 0/2 | 0/4 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 3/11 | 1/4 | 5/7 | 8/8 | 6/8 | 8/8 | 6/6 | 0/2 | 2/6 | 2/6 | 0/4 | 5/5 | 3/4 | 2/2 | 4/4 | 4/4 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 and 2: Placebo (Fasted State) (N=11) | Cohort 1 and 2: Placebo (Fed State) (N=4) | Cohort 1: PF-06954522 Dose Level C (N=7) | Cohort 1: PF-06954522 Dose Level D (N=8) | Cohort 1: PF-06954522 Dose Level D (Fed State High Fat Meal) (N=8) | Cohort 1: PF-06954522 Dose Level E (N=8) | Cohort 1: PF-06954522 Dose Level F (N=6) | Cohort 2: Placebo Standard Meal (N=2) | Cohort 2: PF-06954522 Dose Level A (Fed State-standard Meal) (N=6) | Cohort 2: PF-06954522 Dose Level B (N=6) | Cohort 2: PF-06954522 Dose Level B (Fed State High-fat Meal) (N=4) | Cohort 2: PF-06954522 Dose Level F (N=5) | Cohort 3: Placebo (N=4) | Cohort 3: Placebo (Fed) (N=2) | Cohort 3: PF-06954522 Dose Level D (N=4) | Cohort 3: PF-06954522 Dose Level D (Fed State High-fat Meal) (N=4) | Cohort 3: PF-06954522 Dose Level E (N=3)
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Extraocular muscle disorder (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 3 | 6 | 5 | 4 | 4 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 3 | 3 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 5 | 4 | 7 | 4 | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 4 | 3 | 2
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic enzymes increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine amphetamine positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 1
Food craving (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain fog (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 3 | 3 | 5 | 3 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 4 | 4 | 3
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 1 | 2
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Any untoward findings identified on physical examination and/or cardiac telemetry conducted during the active collection period were captured as adverse events, if those findings met the definition of an AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/77/NCT06003777/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT06003777/SAP_001.pdf